CLINICAL TRIAL: NCT07240285
Title: The Relationship Between Central Sensitization, Pain, and Psychosocial Factors in Individuals With Lipedema: A Cross-Sectional Study
Brief Title: The Relationship Between Central Sensitization, Pain, and Psychosocial Factors in Individuals With Lipedema
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Istftreah
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Lipedema
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lipedema group: Patients with lipedema
- Control group: Patients without lipedema

SUMMARY:
This cross-sectional study will include women aged 18-75 with clinically diagnosed lipedema and healthy controls. Sociodemographic and clinical data will be collected, and participants will complete the Central Sensitization Inventory (CSI), Visual Analog Scale (VAS), Hospital Anxiety and Depression Scale (HADS), and Pain Catastrophizing Scale (PCS). Pain pressure thresholds (PPT) will be assessed using a digital algometer at the middle deltoid, lateral thigh, and medial knee, with three measurements taken at each site and the average recorded.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with lipedema
* Aged between 18 and 75 years
* Provided voluntary informed consent

Exclusion Criteria:

* History of systemic diseases such as diabetes, rheumatologic disorders, or malignancy
* Presence of neurological disorders (e.g., polyneuropathy, multiple sclerosis, history of stroke)
* Currently under active psychiatric treatment Pregnancy
* History of lower extremity surgery or major trauma within the past 6 months
* Received injection therapy or physical therapy for the lower extremities within the past 6 -months
* History of infection or active dermatological disease affecting the lower extremities

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: -Patients with and without lipedema
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-10-10 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Central Sensitization Inventory (CSI) | Baseline
  The CSI assesses symptoms related to central sensitization, such as widespread pain, fatigue, and sleep disturbance. Scores range from 0 to 100, with higher values indicating a greater degree of central sensitization.

SECONDARY OUTCOMES:
Pain Intensity (Visual Analog Scale - VAS) | Baseline
  Pain intensity will be rated on a 10-cm scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores reflect greater perceived pain severity.
Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A): | Baseline
  The HADS-A assesses anxiety symptoms in non-psychiatric populations. Scores range from 0 to 21; higher scores indicate greater anxiety severity.
Hospital Anxiety and Depression Scale - Depression Subscale (HADS-D) | Baseline
  The HADS-D evaluates depressive symptoms, with scores ranging from 0 to 21. Higher scores indicate more severe depressive symptoms.
Pain Catastrophizing Scale (PCS): | Baseline
  he PCS measures negative cognitive and emotional responses to pain. Scores range from 0 to 52, with higher scores indicating greater pain catastrophizing.
Pain Pressure Threshold (PPT): | Baseline
  PPT will be measured using a digital algometer at the middle deltoid, lateral thigh, and medial knee. Lower values indicate greater pain sensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)